CLINICAL TRIAL: NCT05018325
Title: Assessing Effect of Withdrawal Time on Adenoma Detection Rate for Screening Colonoscopy: A Randomized Tandem Study
Brief Title: Assessing Effect of Withdrawal Time on Adenoma Detection Rate for Screening Colonoscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 202103025
Record Dates: First submitted 2021-08-12; First posted 2021-08-24 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Colon Cancer; Rectal Cancer; Colorectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Colonoscopy 6 minute withdrawal time (Active Comparator): -Undergo colonoscopy with the standard 6-minute withdrawal time followed by a tandem colonoscopy of at least another 6-minute withdrawal time.
  Interventions: Procedure: Colonoscopy with 6 minute withdrawal
- Arm 2: Colonoscopy 9 minute withdrawal time (Experimental): -Undergo a 9-minute withdrawal time followed by a tandem colonoscopy with at least the standard 6-minute withdrawal time.
  Interventions: Procedure: Colonoscopy 9 minute withdrawal
- Arm 3: Colonoscopy 12 minute withdrawal time (Experimental): -Undergo colonoscopy with a 12-minute withdrawal time followed by a tandem colonoscopy with at least the standard 6-minute withdrawal time
  Interventions: Procedure: Colonoscopy 12 minute withdrawal

INTERVENTIONS:
Procedure: Colonoscopy with 6 minute withdrawal — Withdrawal time will be determined using a digital stopwatch by the nursing staff.
  Arms: Arm 1: Colonoscopy 6 minute withdrawal time
Procedure: Colonoscopy 9 minute withdrawal — Withdrawal time will be determined using a digital stopwatch by the nursing staff.
  Arms: Arm 2: Colonoscopy 9 minute withdrawal time
Procedure: Colonoscopy 12 minute withdrawal — Withdrawal time will be determined using a digital stopwatch by the nursing staff.
  Arms: Arm 3: Colonoscopy 12 minute withdrawal time

SUMMARY:
The investigators' null hypothesis is that a withdrawal time of 9 to 10 minutes is non-inferior to a withdrawal time of 12 minutes or greater. Thus, the goal of this tandem design trial is to compare the additional diagnostic yield (# of missed lesions) for withdrawal times exceeding 10 minutes for screening/surveillance colonoscopies. Although withdrawal times longer than the standard 6-minute recommendation have been shown to be beneficial, there is limited prospective evidence investigating the benefit or lack thereof for withdrawal times greater than 9-10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 18 and 75 years
* Must be a patient undergoing screening or surveillance colonoscopy
* Must be able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Inability to provide informed consent.
* Personal history of colorectal cancer (CRC)
* Personal history of colon surgery or colon resection
* Personal history of Inflammatory bowel disease
* Personal history of familial polyposis
* Current pregnancy
* Active GI bleeding
* Colonoscopy exams where the cecum cannot be reached (randomization will occur after cecum is reached).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Miss rate of polyps | Time of colonoscopy (day 1)
  * Miss rate = missed polyps/missed polyps + polyps found during 1st exam
  * Polyps is defined as adenomas and sessile serrated adenomas (SSA)

SECONDARY OUTCOMES:
Miss rate of advanced adenomas | Time of colonoscopy (day 1)
  * Miss rate = missed advanced adenomas/missed advanced adenomas + advanced adenomas found during 1st exam
  * Advanced adenoma defined as a polyp ≥ 10mm, adenomas with high-grade dysplasia or villous architecture, serrated lesions with dysplasia, or traditional serrated adenomas

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Kushnir, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported, after deidentification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication without an end date
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu